CLINICAL TRIAL: NCT03847376
Title: Rilpivirine Long Acting Single Patient Requests
Brief Title: Pre-Approval Access to Rilpivirine Long Acting (RPV LA) Injectable Suspension for the Treatment of a Participant With Human Immunodeficiency Virus (HIV)-1 Infection
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Sciences Ireland UC (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108331; TMC278LAHTX2001 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2019-02-18; First posted 2019-02-20 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: HIV
Keywords: Rilpivirine; Long Acting Rilpivirine Injection; HIV; Rilpivirine Expanded Access; Rilpivirine Single Patient Request

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Rilpivirine Long Acting (RPV LA) — Participants will receive RPV LA injectable suspension containing 300 milligram per milliliter (mg/mL) of RPV by intramuscular (IM) injection. A starting dose of 900 milligram (mg) RPV LA (3 milliliter [mL] suspension) will be administered with subsequent doses of 600 mg RPV given at 4-week intervals.
  Other Names: JNJ-16150108-AAA

SUMMARY:
The main purpose of this pre-approval access program (PAAP) is to provide rilpivirine Long Acting (RPV LA) injectable suspension for the treatment of human immunodeficiency virus (HIV)-1 infection as single patient request to individuals who have no available treatment alternatives and/or limited treatment options (for example, who are unable to participate in the Phase III clinical studies or do not qualify). RPV LA can only be provided if participants are also eligible for cabotegravir Long Acting injections.

Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC